CLINICAL TRIAL: NCT01347112
Title: Varenicline Treatment for Active Alcoholic Smokers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivana Croghan, PhD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-008559; 10-008309 (Other: Mayo Clinic IRB # for Grant)
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Smoking; Tobacco Dependence; Alcohol Dependence
Keywords: smoking; tobacco dependence; alcohol dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Alcoholism | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Active Comparator): varenicline 1.0 mg twice daily for 12 weeks
  Interventions: Drug: Varenicline
- Sugar Pil (Placebo Comparator): Varenicline look alike sugar pill twice daily for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Varenicline — varenicline 1.0 mg dose, twice daily for 12 weeks
  Other Names: chantix; champix; varenicline tartrate
  Arms: Varenicline
Drug: placebo — sugar pill twice daily for 12 weeks
  Other Names: sugar pill
  Arms: Sugar Pil

SUMMARY:
Alcohol dependence is a significant and prevalent public health problem affecting approximately 4% of the U.S. adult population. Individuals with alcohol dependence actively seek treatment annually, and long-term alcohol abstinence varies from 40-60%. Because of the high smoking prevalence and trends toward heavier smoking, alcoholic smokers are at high risk for both morbidity and mortality related to alcohol consumption and tobacco dependence. Although several studies have evaluated pharmacotherapy for tobacco dependence in recovering alcoholic smokers, few have evaluated pharmacotherapy for tobacco dependence among currently drinking alcoholic smokers.

Varenicline is the most effective medication currently available for treating tobacco dependence. While some randomized trials have included recovering alcoholics, active alcoholism has been an exclusion criteria for these trials. Thus, this proposal would be the first such clinical trial in currently drinking alcoholic smokers. In addition to helping smokers to stop smoking, varenicline has also been shown to reduce alcohol consumption in rats. The goal of this proposal is to explore the potential efficacy of varenicline for treating tobacco dependence and reducing drinking among alcohol dependent smokers.

The investigators hypothesize that 12 weeks of treatment with varenicline, a partial nicotinic acetylcholine receptor agonist will be more effective than placebo in treating tobacco dependence and reducing nicotine withdrawal symptoms in currently drinking alcoholic smokers. The investigators will also explore whether varenicline has an effect on drinking behavior among currently drinking alcoholics. The investigators propose the following specific aims to test these hypotheses in 70 currently drinking alcoholic smokers recruited at the Mayo Clinic in Rochester, Minnesota.

DETAILED DESCRIPTION:
Seventy smokers who are currently alcohol dependent will be enrolled to this study. If found to be study eligible they will be randomized to either active varenicline or placebo for 12 weeks. During these two weeks, they will be seen either weekly or biweekly. At the end of treatment, they will be followed up for an addition 12 weeks. Their last study visit will be 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female cigarette smokers 18-years-of-age or older and reporting smoking at least an average of 10 cigarettes per day for the past year;
2. Subject is alcohol dependence based on DSM IV criteria as assessed by the Mini-International Neuropsychiatric Interview (MINI) and the physician investigator;3
3. Subject is currently drinking alcoholic beverages as assessed by the physician investigator;
4. Subject is a female subject of non-childbearing potential or a female subject of childbearing potential - who is using contraceptives and has a negative pregnancy test result;
5. Subject must be able to complete all the study visits;
6. Subject has the ability to participate fully in all aspects of the study and keep scheduled appointments;
7. Subject must be in good general health as determined by medical history, physical exam and physician investigator;
8. Subject must provide written informed consent to participate in the study;

Exclusion Criteria:

1. Subject is a female who is pregnant, lactating or likely to become pregnant during the trial and not willing to use an acceptable form of contraception during the medication phase, (for women of child-bearing potential, a pregnancy test will be performed prior to entry into the study and at the end of the medication phase);
2. Subject has another household member in study;
3. Known allergy to varenicline;
4. Subject is currently (in previous 30 days) using other behavioral or pharmacologic tobacco cessation program (i.e., behavioral therapy, nicotine replacement therapy, clonidine, varenicline, bupropion SR, nortriptyline or doxepin) and unwilling or unable to discontinue use;
5. Subject has an unstable medical condition as determined by the physician investigator;
6. Subject describes having a medical history of: a) unstable angina; b) myocardial infarction within the past 3 months; c) coronary angioplasty or d) an untreated cardiac dysrhythmia;
7. Subject has a personal history of renal failure or is on renal dialysis;
8. Subject has a current moderate or severe depression as assessed by the Center for Epidemiologic Studies-Depression survey (CES-D) and physician investigator;
9. Subject has, as defined by the Columbia Suicide Severity Rating Scale (C-SSRS) current non-specific suicidal thoughts, or have a lifetime history of a suicidal attempt (defined as "potentially self-injurious act committed with at least some wish to die, as a result of act");
10. Subject has current (past 30 days) major depressive disorder or has a history of another psychiatric disorder such as psychosis or bipolar disorder;
11. Subject currently uses of other tobacco products (i.e. pipe, cigar, smokeless tobacco) within the past 30 days;
12. Subject currently has cancer [excluding non melanoma skin cancer] not in remission (cancer free for 5 years or more);
13. Subject currently has Type 1 diabetes;
14. Subject has untreated hypertension or baseline systolic blood pressure > 180 or diastolic > 100;
15. Subject is currently on treatment with another investigational drug (within 30 days of study entry);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Hurt, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Franciscan Skemp Hospital, La Crosse, Wisconsin

REFERENCES:
- [Result] Hurt RT, Ebbert JO, Croghan IT, Schroeder DR, Hurt RD, Hays JT. Varenicline for tobacco-dependence treatment in alcohol-dependent smokers: A randomized controlled trial. Drug Alcohol Depend. 2018 Mar 1;184:12-17. doi: 10.1016/j.drugalcdep.2017.11.017. Epub 2018 Jan 2. PMID 29324248
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: Varenicline for tobacco-dependence treatment in alcohol-dependent — http://doi.org/10.1016/j.drugalcdep.2017.11.017

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Varenicline look alike sugar pill twice daily for 12 weeks
  placebo: sugar pill twice daily for 12 weeks
Period: Overall Study
Arm/Group | Varenicline | Sugar Pill
Started | 16 | 17
Completed | 12 | 5
Not Completed | 4 | 12
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Population: Intention to treat all randomized subjects included in study
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Sugar Pill | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.9) | 38.8 (10.4) | 39.5 (11.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
tobacco use [Mean (Standard Deviation); unit: cigarettes per day] | 19.1 (7.5) | 21.6 (7.3) | 20.4 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Smoking Abstinence at End of 12 Weeks of Varenicline Treatment
Description: Prolonged smoking abstinence will be identified by a negative response to the question, "Since 2 weeks after your TQD, have you smoked any tobacco, even a puff, for 7 consecutive days or at least once each week on 2 consecutive weeks?"
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Sugar Pil
Number analyzed (Participants) | 16 | 17
participants | 6 | 1
Statistical Analysis 1: Comparison: Varenicline vs Sugar Pil; Test type: Superiority or Other; p = 0.034, Fisher Exact — 1 tailed fisher's exact test; 1 tailed

2. Secondary Outcome: Prolonged Abstinence at 24 Weeks
Description: Prolonged abstinence is identified by a negative response to the question, "Since 2 weeks after your TQD, have you smoked any tobacco, even a puff, for 7 consecutive days or at least once each week on 2 consecutive weeks?"
Time Frame: week 24
Measure: Number; unit: participants
Arm/Group | Varenicline | Sugar Pil
Number analyzed (Participants) | 16 | 17
participants | 4 | 0
Statistical Analysis 1: Comparison: Varenicline vs Sugar Pil; Test type: Superiority or Other; p = 0.044, Fisher Exact — 1 tailed fisher's exact; 1 tailed

3. Secondary Outcome: Heavy Drinking Days at End of Treatment
Description: Heavy drinking is defined as 5 standard alcohol drinks or greater for men and 4 standard alcohol drinks or greater for women. The number of heavy drinking days per month was determined using the timeline follow-back method.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Varenicline | Sugar Pill
Number analyzed (Participants) | 16 | 17
days | 7.9 (8.3) | 9.1 (7.2)
Statistical Analysis 1: Comparison: Varenicline vs Sugar Pill; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3, 90% CI 2-sided [-4.7 to 2.1] — data were analyzed using analysis of covariance with treatment as the independent variable and the baseline value included as the co-variate

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Varenicline | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 5/16 | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=16) | Sugar Pill (N=17)
nausea (Gastrointestinal disorders) | 4 | 0
sleep disturbance (General disorders) | 2 | 0
vivid dreams (General disorders) | 1 | 1
depressed mood (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes